CLINICAL TRIAL: NCT06071494
Title: A Randomized Controlled Trial Of The Effect Of Tropical Fruits On Intraocular Pressure And Retinal Nerve Fibre Layer Thickness In Patients With Primary Glaucoma
Brief Title: The Effect Of Tropical Fruits In Patients With Primary Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, NURUL MUNIRAH BINTI MOHAMAD, Principle Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RSCH ID-23-03744-7U6
Record Dates: First submitted 2023-10-01; First posted 2023-10-06 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Primary Glaucoma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tropical Fruits (Experimental): patient will be consuming the chosen fruits, according to the size of the serving following Malaysian Dietary Guideline 2020
  Interventions: Other: Tropical fruits
- Normal diet (No Intervention): patient will consume normal diet as usual

INTERVENTIONS:
Other: Tropical fruits — papaya, mango, banana, orange
  Arms: Tropical Fruits

SUMMARY:
To evaluate the effect of regular tropical fruits intake in primary glaucoma patients.

Methodology :

Research Design Randomized controlled trial

Study Duration February 2024-June 2025

Study Location

1. Ophthalmology Clinic, Hospital Universiti Sains Malaysia, Kelantan

Source Reference Population Adults with primary glaucoma in Peninsular Malaysia

Study Source Population Adults with primary glaucoma attending Ophthalmology clinic, Hospital Universiti Sains Malaysia during study duration.

DETAILED DESCRIPTION:
General objective To evaluate the effect of regular tropical fruits intake on intra-ocular pressure (IOP) and retinal nerve fibre layer thickness (RNFL) in primary glaucoma patients.

Research hypothesis

1. There is a significant different in the IOP measurement between those whose taking regular tropical fruits and not taking them at baseline, 1 month, 3 month and 6 month among patients with primary glaucoma.
2. There is a significant different in RNFL thickness between those whose taking regular tropical fruits and not taking them at baseline, 1 month, 3 month and 6 month among patients with primary glaucoma.

Inclusion Criteria

1. Patient with confirmed diagnosis of POAG and PACG
2. Patient on medical treatment and achieved target IOP in last 6 months
3. Good compliance with pressure lowering agents

Exclusion Criteria

1. Poorly controlled diabetes mellitus, hypertension and hyperlipidaemia
2. Active smoker
3. Mentally challenge based on diagnosis
4. History of previous intraocular surgery other than uncomplicated cataract surgery within past 6 months
5. Poor signal strength OCT RNFL
6. Patient with media opacities that affect the reliability of OCT measurements , such as Cornea opacity, dense cataract with LOCS III of more than grade 2, vitreous haemorrhage
7. Other optic neuropathy apart from glaucoma
8. History of taking antioxidant supplement 3 months prior to recruitment.

Methods of Data Collection

This study will be conducted after obtaining ethical approval from the Universiti Sains Malaysia Ethical Committee (JPeM) and will be conducted in accordance to World Medical Association Declaration of Helsinki ethical principles for medical research involving human subjects.

Recruitment of Subject

Patient diagnosed with POAG and PACG attending Ophthalmology clinic, Hospital USM during study duration and fulfilled study inclusion and exclusion criteria. An informed and written consent will be taken and information form given to patients. The selected patients will be randomized into 2 groups (A and B) using sequentially numbered, opaque sealed envelopes (SNOSE). Group A patient will be consuming the chosen fruits and group B patient will not consume them.

Interventional Protocol

Patients in Group A will have to consume 2 types of fresh fruits per week as 2 servings once per day, daily for a 6-month duration. The chosen fruits are papaya, banana, mango and orange, and 2 types of fruits per week will be determined by the primary investigator. Size of the servings is according to the Malaysian Dietary Guideline 2020. They must eat them raw, and not to process or cook them in any other way. The fruits will be distributed by research assistant weekly throughout the study period. Patient will be reminded weekly using text messages or phone call by a research assistant for the fruit's consumption. Patients in group A and group B will be given a dietary diary throughout the study period, where the patient will mark the intake of fruits listed. The purpose of the diary is also to monitor patient intake of the fruits and daily diet as well.

IOP measurement

IOP measurement will be done using Goldmann Applanation Tonometer (GAT) in sitting position by the primary investigator (Nurul Munirah) who will be blinded. GAT will be calibrated daily before use to measure the IOP. Measurement of IOP will be done only at 8am - 10am (to prevent diurnal variation). Before IOP measurement, subjects are advised to avoid drinking coffee or any caffeinated drink 24 hours before and only to take light meal 2 hours before (to reduce the effect of hyperglycaemia and hydration on IOP). Only one eye will be measured, if both eyes are eligible, only right eye will be selected regardless of severity of glaucoma. Three readings of IOP will be measured and the mean reading will be taken as result. IOP measurement will be taken at baseline, first, third and sixth month post recruitment for group A and B.

OCT evaluation on RNFL thickness

Spectral domain Cirrus HD-OCT will be used to measure RNFL thickness and ONH parameters by a trained personnel who is blinded. Patient's eye will be dilated and patient will sit and rest his/her head on a support to keep it motionless in front of the OCT machine. The OCT will then scan patient's eye without touching it. Scans with signal strength less than 6, eye movement or blinking artifacts within the 1.73-mm radius around the ONH, or with segmentation errors will be repeated. If there is unsatisfactory measurement after 3 attempts, the patient will be excluded from the study. OCT will be conducted at baseline, first, third and sixth month post recruitment for group A and B.

Data Entry and Statistical Analysis

The data entry and analysis will be performed by using Statistical Package for the Social Sciences (SPSS) version 29 licensed to USM.

* Paired T-test
* Chi-square test
* A one-way repeated measures analysis of variance (RM ANOVA)

Plans for minimizing study errors

These steps will be taken to minimize the errors while conducting the study:

* The same instruments and equipment will be used for repeated measurement in this study.
* The measurement of IOP will be done at the same time (8am-10am) in a day for all patients (to prevent diurnal variation).
* OCT measurements will be performed by qualified and trained personnel only.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with confirmed diagnosis of POAG and PACG
2. Patient on medical treatment and achieved target IOP in last 6 months
3. Good compliance with pressure lowering agents

Exclusion Criteria:

1. Poorly controlled diabetes mellitus, hypertension and hyperlipidaemia
2. Active smoker
3. Mentally challenge based on diagnosis
4. History of previous intraocular surgery other than uncomplicated cataract surgery within past 6 months
5. Poor signal strength OCT RNFL
6. Patient with media opacities that affect the reliability of OCT measurements , such as Cornea opacity, dense cataract with LOCS III of more than grade 2, vitreous haemorrhage
7. Other optic neuropathy apart from glaucoma
8. History of taking antioxidant supplement 3 months prior to recruitment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
intraocular pressure | baseline, at 1 month , at 3 months and 6 months
  tonometer
retinal nerve fibre layer | baseline, at 1 month , at 3 months and 6 months
  Spectral domain Cirrus HD-OCT

CONTACTS AND LOCATIONS:
Overall Officials: Nurul Munirah Mohamad, Dr, Principal Investigator — Department of Ophthalmology School of Medical Sciences Universiti Sains Malaysia,Health Campus.; Liza Sharmini Ahmad Tajudin, Prof. Dr., Study Chair — Department of Ophthalmology School of Medical Sciences Universiti Sains Malaysia,Health Campus.; Rohana Abd Jalil, Ass. Prof., Study Director — Department of Ophthalmology School of Medical Sciences Universiti Sains Malaysia,Health Campus.; Fatimah Suhaila Sukaimy, Dr, Study Director — Department of Ophthalmology Hospital Tengku Ampuan Afzan, Ministry of Health, Malaysia
Locations (1):
- Univerisiti Sains Malaysia, Kubang Kerian, Kota Bharu, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weinreb RN, Khaw PT. Primary open-angle glaucoma. Lancet. 2004 May 22;363(9422):1711-20. doi: 10.1016/S0140-6736(04)16257-0. PMID 15158634
- [Background] Braakhuis A, Raman R, Vaghefi E. The Association between Dietary Intake of Antioxidants and Ocular Disease. Diseases. 2017 Jan 30;5(1):3. doi: 10.3390/diseases5010003. PMID 28933356
- [Background] Kang JH, Willett WC, Rosner BA, Buys E, Wiggs JL, Pasquale LR. Association of Dietary Nitrate Intake With Primary Open-Angle Glaucoma: A Prospective Analysis From the Nurses' Health Study and Health Professionals Follow-up Study. JAMA Ophthalmol. 2016 Mar;134(3):294-303. doi: 10.1001/jamaophthalmol.2015.5601. PMID 26767881
- [Background] Neufeld AH, Sawada A, Becker B. Inhibition of nitric-oxide synthase 2 by aminoguanidine provides neuroprotection of retinal ganglion cells in a rat model of chronic glaucoma. Proc Natl Acad Sci U S A. 1999 Aug 17;96(17):9944-8. doi: 10.1073/pnas.96.17.9944. PMID 10449799
- See also: Primary open-angle glaucoma — https://pubmed.ncbi.nlm.nih.gov/15158634/
- See also: The Association between Dietary Intake of Antioxidants and Ocular Disease. Diseases — https://pubmed.ncbi.nlm.nih.gov/28933356/
- See also: Association of Dietary Nitrate Intake With Primary Open-Angle Glaucoma: A Prospective Analysis From the Nurses' Health Study and Health Professionals Follow-up Study — https://pubmed.ncbi.nlm.nih.gov/26767881/
- See also: Inhibition of nitric-oxide synthase 2 by aminoguanidine provides neuroprotection of retinal ganglion cells in a rat model of chronic glaucoma — https://pubmed.ncbi.nlm.nih.gov/10449799/